CLINICAL TRIAL: NCT04188405
Title: A Phase II Study of the Combination of Decitabine, Venetoclax, and Ponatinib in Patients With Philadelphia Chromosome-Positive Acute Myeloid Leukemia or Myeloid Blast Phase Chronic Myelogenous Leukemia
Brief Title: Decitabine, Venetoclax, and Ponatinib for the Treatment of Philadelphia Chromosome-Positive Acute Myeloid Leukemia or Myeloid Blast Phase or Accelerated Phase Chronic Myelogenous Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0610; NCI-2019-07594 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0610 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-25; First posted 2019-12-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Myeloid Leukemia; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Acute Myeloid Leukemia; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Acute; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Decitabine; Injections; ponatinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ponatinib, venetoclax, decitabine) (Experimental): See Detailed Description.
  Interventions: Drug: Decitabine; Drug: Ponatinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Ponatinib — Given PO
  Other Names: AP-24534; AP24534
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well the combination of decitabine, venetoclax, and ponatinib work for the treatment of Philadelphia chromosome-positive acute myeloid leukemia or myeloid blast phase or accelerated phase chronic myelogenous leukemia. Drugs used in chemotherapy such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Ponatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving decitabine, venetoclax, and ponatinib may help to control Philadelphia chromosome-positive acute myeloid leukemia or myeloid blast phase or accelerated phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of the regimen, as defined by the rate of complete remission (CR) or CR with incomplete count recovery (CRi).

SECONDARY OBJECTIVES:

I. To determine efficacy outcomes, including rate of minimal residual disease negativity by flow cytometry and polymerase chain reaction (PCR) for BCR-ABL1 transcripts, median relapse-free survival, and median overall survival.

II. To determine the proportion of patients proceeding to allogeneic stem cell transplant (ASCT).

III. To preliminarily determine the safety of the combination regimen.

EXPLORATORY OBJECTIVES:

I. To evaluate the effect of single-agent ponatinib on apoptotic proteins and Bcl-2 dependency.

II. To correlate apoptotic protein expression and Bcl-2 dependency on response and resistance to the combination regimen.

OUTLINE:

Patients recently (within 2 weeks of anticipated start date) treated with ponatinib receive ponatinib orally (PO) daily on days 1-21 of cycle 1 and days 1-28 of subsequent cycles, venetoclax PO daily on days 1-21, and decitabine intravenously (IV) over 60 minutes on days 1-5. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients who have not been recently (within 2 weeks of anticipated start date) treated with ponatinib may receive ponatinib monotherapy PO daily on days 1-7 before starting combination therapy with venetoclax in cycle 1. After completion of ponatinib lead-in, patients will receive ponatinib PO daily on days 1-21 of cycle 1 and on days 1-28 of subsequent cycles, venetoclax PO daily on days 8-28 of cycle 1 and days 1-21 of subsequent cycles, and decitabine IV over 60 minutes on days 8-12 of cycle 1 and days 1-5 of subsequent cycles. For these patients, cycle 1 is 35 days in duration and cycles 2-24 repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Philadelphia (Ph)+ acute myeloid leukemia (AML) or myeloid accelerated phase (AP)-chronic myelogenous leukemia (CML) or blast phase (BP)-CML (either t[9;22] and/or BCR-ABL1 positive by fluorescent in situ hybridization or polymerase chain reaction). Both untreated and relapsed/refractory patients are eligible
* Performance status =< 3 (Eastern Cooperative Oncology Group [ECOG] scale)
* Total serum bilirubin =< 2 x upper limit of normal (ULN), unless due to Gilbert's syndrome, hemolysis or the underlying leukemia approved by the principal investigator (PI)
* Alanine aminotransferase (ALT) =< 1.5 x ULN, unless due to the underlying leukemia approved by the PI
* Aspartate aminotransferase (AST) =< 1.5 x ULN unless due to the underlying leukemia approved by the PI
* Creatinine clearance >= 30 mL/min
* Serum lipase =< 1.5 x ULN
* Amylase =< 1.5 x ULN
* Ability to swallow
* Signed informed consent

Exclusion Criteria:

* Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of improvement despite antimicrobial treatment)
* History of acute pancreatitis within 6 months of study or history of chronic pancreatitis
* Uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL)
* Active secondary malignancy that in the investigator's opinion will shorten survival to less than 1 year
* Active grade III-V cardiac failure as defined by the New York Heart Association criteria
* Clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

  * Myocardial infarction (MI), stroke, revascularization, unstable angina or transient ischemic attack within 6 months
  * Left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards prior to enrollment
  * Diagnosed or suspected congenital long QT syndrome
  * Clinically significant atrial or ventricular arrhythmias (such as uncontrolled, clinically significant atrial fibrillation, ventricular tachycardia, ventricular fibrillation, or torsades de pointes) as determined by the treating physician
  * Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 480 msec) unless corrected after electrolyte replacement
  * History of venous thromboembolism including deep venous thrombosis or pulmonary embolism within the past 3 months, excluding line-associated deep venous thrombosis (DVT) of the upper extremity
  * Uncontrolled hypertension (diastolic blood pressure > 100 mmHg; systolic > 150 mmHg)
* Consumed grapefruit, grapefruit products, Seville oranges, or star fruit within 3 days prior to starting venetoclax
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator. Prior recent treatment with corticosteroids, hydroxyurea, or a Food and Drug Administration (FDA)-approved BCR-ABL tyrosine kinase inhibitor (TKI) is permitted
* Pregnant and lactating women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception throughout the study period. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | End of cycle 2 (each cycle is 28 days)
  Defined as the proportion of patients achieving complete remission (CR) + CR with incomplete count recovery (CRi) occurring at the end of 2 cycles of treatment. Will be estimated along with the 95% credible interval. Patients who drop out of the study before completing 2 cycles and have been treated will be censored for the primary endpoint analysis.

SECONDARY OUTCOMES:
Rate of minimal residual disease negativity | Up to 4.5 years
  Will be estimated along with the 95% credible interval.
Proportion of patients proceeding to allogeneic stem cell transplant | Up to 4.5 years
  Will be estimated along with the 95% credible interval.
Relapse-free survival (RFS) | From the date of treatment initiation to the date of documented treatment relapses from CR/CRi or death from any cause, whichever occurs first, assessed up to 4.5 years
  The distribution of RFS will be estimated using the method of Kaplan and Meier. Comparisons by important subgroups will be made using the log-rank tests.
Overall survival (OS) | From treatment start till death or last follow-up, assessed up to 4.5 years
  The distribution of OS will be estimated using the method of Kaplan and Meier. Comparisons by important subgroups will be made using the log-rank tests.
Incidence of adverse events | Up to 4.5 years
  Safety data will be summarized by category, severity and frequency.

OTHER OUTCOMES:
Apoptotic protein expression and Bcl-2 dependency on response and resistance | Up to 4.5 years
  The association between response and patient's clinical information such as apoptotic protein expression, etc. will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Short, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Short NJ, Nguyen D, Jabbour E, Senapati J, Zeng Z, Issa GC, Abbas H, Nasnas C, Qiao W, Huang X, Borthakur G, Chien K, Haddad FG, Pemmaraju N, Karrar OS, Nguyen D, Konopleva M, Kantarjian H, Ravandi F. Decitabine, venetoclax, and ponatinib for advanced phase chronic myeloid leukaemia and Philadelphia chromosome-positive acute myeloid leukaemia: a single-arm, single-centre phase 2 trial. Lancet Haematol. 2024 Nov;11(11):e839-e849. doi: 10.1016/S2352-3026(24)00250-3. Epub 2024 Sep 17. PMID 39303729
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT04188405/ICF_000.pdf